CLINICAL TRIAL: NCT03202459
Title: Prophylaxy of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Lígia Andrade da Silva Telles mathias, Doctor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 56057116.0.0000.5479
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Complications; Postoperative Nausea and Vomiting
Keywords: Anesthesia; Complications; Nausea; Vomiting
MeSH Terms: conditions — Postoperative Complications; Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: Group A - gabapentin (Active Comparator): The patient will receive oral 600 mg gabapentin 2 h before surgery
  Interventions: Drug: Group A - gabapentin 600 mg
- Active Comparator: Group B - pregabalin (Active Comparator): The patient will receive oral pregabalin 150 mg 2 h before surgery
  Interventions: Drug: Group B - pregabalin
- Placebo Comparator: Group C - placebo (Placebo Comparator): The patient will receive oral placebo 2 h before surgery and ondansetron 8mg intravenous at the end of the surgery
  Interventions: Drug: Group C - placebo

INTERVENTIONS:
Drug: Group A - gabapentin 600 mg — The patient will receive oral 600 mg gabapentin 2 h before surgery
  Arms: Active Comparator: Group A - gabapentin
Drug: Group B - pregabalin — The patient will receive oral pregabalin 150 mg 2 h before surgery
  Arms: Active Comparator: Group B - pregabalin
Drug: Group C - placebo — The patient will receive oral placebo 2 h before surgery and ondansetron 8mg intravenous at the end of the surgery
  Arms: Placebo Comparator: Group C - placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) is one of the most commonly reported adverse effects of anesthesia. The general incidence of vomiting is approximately 30%, nausea at 50% and the PONV rate can go up to 80% in high-risk patients without prophylaxis. Prevention of these episodes in high-risk patients improves satisfaction and well-being rates. Therefore, it becomes important the adequate control of PONV, aiming at the satisfaction of the patient with the procedure, lower costs for the health system as well as reduction of complications in the postoperative period. This study aims to evaluate the association of gabapentin or pregabalin with dexamethasone in reducing the incidence of PONV in high-risk patients undergoing laparoscopic surgeries in the first 48 hours postoperatively as well as to assess side effects.

DETAILED DESCRIPTION:
The study included 60 patients at high risk for PONV (Apfel-score 0, I, II, III and IV) scheduled for elective laparoscopic surgeries at the Central Surgical Center of Irmandade da Santa Casa de Misericórdia in São Paulo. Inclusion criteria will be ASA I or II of either sex, in the age range of 18 to 70 years. In this study, the recruited patients will be allocated randomly into three groups. The group A will receive oral 600 mg gabapentin 2 h before surgery. The group B will receive oral 150 mg pregabalin 2 h before surgery. The Group C will receive oral placebo 2 h before surgery and ondansetron 8mg intravenous at the end of the surgery. This study is "double-blind", in which neither the doctor nor the patient knows what medicine is being given.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic procedures
* Apfel Score 0, I, II, III and IV
* ASA I / II

Exclusion Criteria:

* Patients with surgery converted to open before thirty minutes of surgery
* Patients who were exposed previously to gabapentin or pregabalin Patients who have allergy to any medicine used in the study
* Patient who have to any cognitive impairment
* Illiterate patients
* Patients who refuse to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Nausea or vomiting M0 | 1 hours
  The occurrence of postoperative nausea or vomiting, in the recovery room, during the first hour after surgery
Postoperative Nausea or vomiting M12 | 12 hours
  The occurrence of postoperative nausea or vomiting, reported by the patient or witnessed by a healthcare provider during the first 12 hours after surgery
Postoperative Nausea or vomiting M24 | 24 hours
  The occurrence of postoperative nausea or vomiting, reported by the patient or witnessed by a healthcare provider during the first 24 hours after surgery
Postoperative Nausea or vomiting M48 | 48 hours
  The occurrence of postoperative nausea or vomiting, reported by the patient or witnessed by a healthcare provider during the first 48 hours after surgery

SECONDARY OUTCOMES:
Patient demographic data | Before surgery
  With a questionnaire will be studied the variables: age, sex, weight, height, BMI
Surgical Duration | First hour after surgery
  Time of surgery
Duration of postoperative anesthesia stay | First hours after surgery
  Time to postoperative anesthesia care unit discharge alive (hours)
The length of stay in hospital | From end of surgery until hospital discharge or 30 days after surgery
  Time of stay in hospital
Time to request the first medication for nausea and vomiting | First hour after surgery
  Reported by the patient or by a healthcare provider
Amount of medication | During the first 30 days after surgery
  Reported by a healthcare provider
Postoperative complications | During the first 30 days after surgery
  Postoperative complications after surgery
Degree of patient satisfaction | Before discharge
  The patient's overall satisfaction will be assessed using point scales (very satisfied, somewhat satisfied, neither satisfied nor dissatisfied, somewhat dissatisfied, very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Result] Pandey CK, Priye S, Ambesh SP, Singh S, Singh U, Singh PK. Prophylactic gabapentin for prevention of postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy: a randomized, double-blind, placebo-controlled study. J Postgrad Med. 2006 Apr-Jun;52(2):97-100. PMID 16679671
- [Result] Grant MC, Lee H, Page AJ, Hobson D, Wick E, Wu CL. The Effect of Preoperative Gabapentin on Postoperative Nausea and Vomiting: A Meta-Analysis. Anesth Analg. 2016 Apr;122(4):976-85. doi: 10.1213/ANE.0000000000001120. PMID 26991615
- [Result] Chandrakantan A, Glass PS. Multimodal therapies for postoperative nausea and vomiting, and pain. Br J Anaesth. 2011 Dec;107 Suppl 1:i27-40. doi: 10.1093/bja/aer358. PMID 22156268